CLINICAL TRIAL: NCT06996990
Title: The Relationship Between Injury Risk and Pain, Fatigue, Muscle Strength, Balance and Quality of Life in Volleyball Players
Brief Title: Injury Risk Factors in Volleyball Players
Status: Not yet recruiting | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Principal Investigator, Izmir Democracy University
Other Study IDs: Volleyball players and injury
Record Dates: First submitted 2025-05-16; First posted 2025-05-30 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Injury;Sports; Athletic Injuries
Keywords: Pain; Fatigue; Muscle Strength; Balance; Quality of Life; Volleyball; Sport Injury
MeSH Terms: conditions — Athletic Injuries; Pain; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volleyball Players: This group will consist of active volleyball players competing at a regional or national level. Participants will undergo one-time assessments including muscle strength, balance, fatigue, pain levels, and quality of life.
  Interventions: Other: Physical evaluations in Volleyball Players

INTERVENTIONS:
Other: Physical evaluations in Volleyball Players — This study will evaluate pain, fatigue, muscle strength, balance and quality of life in volleyball players. All these measurements will be completed in two sessions lasting 45-60 minutes.

SUMMARY:
The aim of this study is to examine the relationship between injury risk and pain, fatigue, muscle strength, balance and quality of life in volleyball players. In this context, it will be investigated how the pain and fatigue levels experienced by volleyball players interact with muscle strength and balance and how these factors increase the risk of injury.

DETAILED DESCRIPTION:
Musculoskeletal injuries are highly prevalent among volleyball players and this may be due to the interaction of various physical and subjective factors. Although some risk factors such as muscle strength and balance have been previously investigated, there is limited data on how these parameters together relate to injury risk and athlete health. In this cross-sectional study, standardized tests and self-report questionnaires will be administered to a sample of competitive volleyball players.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old and volunteer
* Have not had any upper or lower extremity injuries in the last 3 months
* Have not had any upper or lower extremity surgery in the last 6 months
* Play volleyball professionally

Exclusion Criteria:

* Having had a lower or upper extremity injury in the last 3 months
* Having had upper or lower extremity surgery in the last 6 months
* Being pregnant

Min Age: 18 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of the research consists of elite athletes and the sample of the research consists of elite volleyball players who volunteered to participate in the research. In our research, there is only one research group consisting of elite volleyball players and there are at least 28 volleyball players.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Injury risc assessment | through study completion, an average of 1 year
  The Functional Movement Screening Test will be used to assess injury risc in athletes. Seven exercises are used in this test. Each movement is scored on a scale from 0 to 3, with a maximum total score of 21. As the score from this test increases, the risk of injury decreases.

SECONDARY OUTCOMES:
Pain intensity evaluation | through study completion, an average of 1 year
  Pain intensity will be assessed using the Numerical Rating Scale, where participants rate their pain intensity from 0 (no pain) to 10 (maximum pain).
Fatigue assessment | through study completion, an average of 1 year
  The Perceived Physical and Cognitive Fatigue Scale will be used to assess athletes' physical and cognitive fatigue. The scale has 19 items, scored ranging from 19 to 95. Higher scores indicate increased perceived fatigue levels.
Forced vital capacity (FVC) | through study completion, an average of 1 year
  Forced vital capacity (FVC) will be evaluated with a spirometer.
Forced expiratory volume in the first second (FEV1) | through study completion, an average of 1 year
  Forced expiratory volume in the first second (FEV1) will be evaluated with a spirometer.
FEV1/FVC | through study completion, an average of 1 year
  FEV1/FVC will be evaluated with a spirometer.
Flow rate 25-75% of forced expiratory volume (FEF 25-75%) | through study completion, an average of 1 year
  Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) will be evaluated with a spirometer.
Peak flow rate (PEF) | through study completion, an average of 1 year
  Peak flow rate (PEF) will be evaluated with a spirometer.
Muscle Strength Measurement | through study completion, an average of 1 year
  The lower extremity muscle strength of athletes will be assessed using isokinetic test. Each maximal voluntary contraction will involve the athlete contracting as hard and as fast as possible from full extension to full flexion.Higher values indicate better muscle strength.
Hand Grip Strength measurement | through study completion, an average of 1 year
  Hand grip strength will be assessed using a hand dynamometer. Participants will perform three trials on each hand . The maximum grip strength value for each hand will be analysed.
Respiratory Muscle Strength measurement | through study completion, an average of 1 year
  Respiratory muscle strength will be evaluated using a spirometer. Athletes will perform maximal inspiration (Müller maneuver) and expiration (Valsalva maneuver) to obtain measurements. The highest value will be used for analysis.
Cough force measurement | through study completion, an average of 1 year
  Cough force will be assessed using a peak flow meter. The highest value of three attempts will be recorded. The high value obtained indicates good cough strength.
Balance evaluation | through study completion, an average of 1 year
  Balance will be assessed using the Y-Balance Test, and the average distance reached will be recorded.
Quality of Life (SF-36 or WHOQOL-BREF) | through study completion, an average of 1 year
  The Short Form-36 (SF-36) will be used to assess quality of life. total score is scored from 0 (poorest health) to 100 (best health), with higher scores indicating better health status.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, Assoc Prof, Study Director — Izmir Democracy University; Rümeysa Binici, PT, Principal Investigator — Aras KArgo Volleyball Club; Güfat Arslan, MD, Principal Investigator — Izmir City Hospital; Uygar Kaya, PT, Principal Investigator — Göztepe Volleyball Club
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soylu, Ç., Altundağ, E., Akarçeşme, C., & Ün Yildirim, N. (2020). The relationship between isokinetic knee flexion and extension muscle strength, jump performance, dynamic balance and injury risk in female volleyball players.
- [Background] Wilkosz P, Kabacinski J, Mackala K, Murawa M, Ostarello J, Rzepnicka A, Szczesny L, Fryzowicz A, Maczynski J, Dworak LB. Isokinetic and Isometric Assessment of the Knee Joint Extensors and Flexors of Professional Volleyball Players. Int J Environ Res Public Health. 2021 Jun 24;18(13):6780. doi: 10.3390/ijerph18136780. PMID 34202540